CLINICAL TRIAL: NCT02565407
Title: Robot-aided Proprioceptive Rehabilitation Training With Additional Vibro-tactile Feedback
Brief Title: Robot-aided Proprioceptive Rehabilitation Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1505M72302
Record Dates: First submitted 2015-08-27; First posted 2015-10-01 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Stroke; Peripheral Sensory Neuropathy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proprioceptive training (Experimental): This arm will receive specialized robot-aided proprioceptive training of the wrist next to usual care.
  Interventions: Behavioral: Proprioceptive training
- Usual care (Active Comparator): This arm will receive what participants have been receiving from their healthcare providers. It may range from no treatment to various sessions of occupational and physical therapy at home, day rehabilitation, or outpatient visits.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Proprioceptive training — Training includes a virtual balance board and center-out task. Small vibratory motors placed on forearms provide vibro-tactile movement feedback (VTF). During familiarization participants learn to associate VTF with wrist movement and visual feedback. Vision is occluded after this phase. In the virtual balance board task participants use wrist motion to roll a ball to a target on the board. VTF indicates the desired movement direction and ball velocity. The center-out task involves wrist motion to control a cursor to reach a target. The wrist robot delivers an assistive force towards the target. VTF signals magnitude and direction of the cursor deviating away from the desired path.
  Arms: Proprioceptive training
Behavioral: Usual care — Usual care refers to care that participants receive through their healthcare providers. It may range from no treatment to various sessions of occupational and physical therapy received at in- or outpatient rehabilitation clinics or at home.
  Arms: Usual care

SUMMARY:
This study investigates the effect of a robot-aided 2-day proprioceptive training of the wrist on the proprioceptive and motor function of the wrist/hand complex in patients with proprioceptive impairment. The wrist proprioceptive training consists of active movement training with augmented haptic and vibro-tactile feedback provided by a patented wrist robotic system (US Serial No. 62/136,065). This study protocol can be applied to a variety of clinical and non-clinical populations. The purpose of this study is to obtain preliminary data on the effectiveness of the proprioceptive training in subjects with cortical stroke or peripheral sensory neuropathy.

DETAILED DESCRIPTION:
This protocol seeks to improve proprioceptive-motor function. Proprioception refers to the perception of limb position or motion and the orientation of one's body in space. Numerous medical conditions with motor symptoms are also associated with proprioceptive loss, such as osteoarthritis, Parkinson's disease, peripheral sensory neuropathy, stroke, and developmental coordination disorder.

However, therapies to improve proprioceptive function in these populations are either non-existent or very limited in scope although it is established that proprioceptive impairments severely degrade motor function. The proposed protocol focuses on proprioception for fine motor function of the hand/wrist joint complex, because hand/wrist motor control is highly important for activities of daily living.

The specific aims are to determine if a 2-day wrist proprioceptive training:

1. improves limb position sense acuity,
2. improves the spatial precision of wrist/hand motor tasks,
3. increases the efficiency of performing such motor tasks,
4. is associated with neural changes in cortical processing as measured by short-latency somatosensory evoke potentials (SEP) and motor evoked potentials (MEP) using transcranial magnetic stimulation.

The study follows a crossover design with two arms and two groups. Time frame for the completion of the study is up to 7 days depending on the start day of the week (Monday through Friday). No testing will occur on the weekend.

Group 1 will have the following time frame: Day 1: pre-test (approx. 3 hrs.) and training intervention (approx. 30 min.). Day 2: training intervention (approx. 30 min.) and post-test 1 (approx. 3 hrs.). Days 3-6: Usual care (min. of 2 days required). Days 5-7: Post-test 2 (depending on the start day of the week, it is either Day 5,6, or 7).

Group 2 will have the following time frame: Day 1: pre-test 1 (approx. 3 hrs.). Days 2-4: Usual care (min. of 2 days required). Days 4-6: pre-test 2 (approx. 3 hrs.) and training intervention (approx. 30 min.). Days 5-7: Training intervention and post-test 1 (depending on the start day of the week, it is either Day 5,6, or 7).

ELIGIBILITY:
For all participants (both healthy and patient populations)

Inclusion Criteria:

1. wrist passive range of motion (ROM) more than 22.5° in flexion/extension
2. sense the vibro-tactile cues on either forearms in order to effectively receive the movement-related feedback
3. resist minimal resistance in gravity-eliminated position (score at least 2+/5 with the physical examination of manual muscle testing (Hislop, Avers, & Brown, 2013)) ) in all wrist movement directions.

Exclusion Criteria:

1. Regular intake of benzodiazepines.
2. Cognitive impairment: score ≥ 23 on Mini-mental state examination (Folstein, Robins & Helzer, 1983)
3. Depressive symptoms: score ≤ 19 on Beck depression inventory (Beck, Steer, & Carbin,1988).

Inclusion Criteria for Stroke Subjects

1. at least 3 months after stroke
2. whose age are between 30 to 75 years old.

Exclusion Criteria for Subjects undergoing the TMS procedure (Rossi, Hallett, Rossini, & Pascual-Leone, 2009)

* Has implanted metal in the body.
* Diagnosed with multiple sclerosis, major psychiatric conditions, epilepsy, history of seizures in the past 2 years, sleep deprivation, pregnancy, uncontrolled migraine, major traumatic head injury, severe heart disease, increased intracranial pressure, high consumption of alcohol, any conditions that predispose one to seizures
* Is currently taking any pro-epileptic medication (e.g. epileptogenic drugs such as tricyclic antidepressants)
* When no electromyography response can be elicited within the range of the TMS stimulator
* Pregnant at the time of data collection .

Ages: 4 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2021-05-24 (Actual)

PRIMARY OUTCOMES:
Joint position sense acuity of the wrist (just-noticeable-difference threshold) | For Group1: Change from pre-test at Day 1 (prior to training) to post-test 1 at Day 2. For Group 2: Change from pre-test 2 at Days 4-6 to post-test 1 at Days 5-7.
  Using the wrist robot, the just-noticeable-difference threshold (JND) of wrist position will measured by a 2-alternative forced choice psychophysical paradigm. Participant's wrist will be passively flexed to two positions (the standard stimulus and the comparison stimuli) in random order. The standard stimulus is always 15° wrist flexion from neutral wrist position and the comparison stimulus is always larger than the standard. Participants indicate verbally which stimulus was perceived as having a larger amplitude. Unit is degrees.

SECONDARY OUTCOMES:
Root-mean-square tracing error as a measure of movement accuracy | For Group1: Change from pre-test at Day 1 (prior to training) to post-test 1 at Day 2. For Group 2: Change from pre-test 2 at Days 4-6 to post-test 1 at Days 5-7.
  Using the wrist robot, participants perform wrist movements to move a cursor on a screen. Task is to trace various template wave forms (saw tooth, sine wave, irregular, figure-of eight) displayed on the screen. The same procedure will be performed with a pen stylus on a digital tablet. The cursor position will be recorded continuously through the tracking task. Root-mean-square tracing error is calculated based on the difference between the cursor path and the template waveform. Unit is in mm.
Movement time | For Group1: Change from pre-test at Day 1 (prior to training) to post-test 1 at Day 2. For Group 2: Change from pre-test 2 at Days 4-6 to post-test 1 at Days 5-7.
  Movement time is the time it takes to complete either the tracing or pointing task. Unit is in seconds.
Jerk cost as a measure of movement smoothness | For Group1: Change from pre-test at Day 1 (prior to training) to post-test 1 at Day 2. For Group 2: Change from pre-test 2 at Days 4-6 to post-test 1 at Days 5-7.
  The jerk cost is defined as the integral of the first derivative of acceleration.
Fugl-Meyer Assessment score | For Group1: Change from pre-test at Day 1 (prior to training) to post-test 1 at Day 2. For Group 2: Change from pre-test 2 at Days 4-6 to post-test 1 at Days 5-7.
  Fugl-Meyer Assessment is a clinical instrument used to evaluate and measure recovery in post-stroke patients. Only the motor section for the upper extremity of the assessment is used (Fugl-Meyer et al., 1974). Range of possible scores is 0 [no recovery] - 66 [full recovery].
Nottingham Sensory Assessment score | For Group1: Change from pre-test at Day 1 (prior to training) to post-test 1 at Day 2. For Group 2: Change from pre-test 2 at Days 4-6 to post-test 1 at Days 5-7.
  Erasmus-modified Nottingham Sensory Assessment is a clinical instrument to evaluate somatosensory function. For this study only the proprioception section of upper limb is used (Stolk-Hornsveld, Crow, Hendriks, Van Der Baan, & Harmeling-Van Der Wel, 2006). Range of possible scores is 0 [absent] - 2 [intact].
Canadian Occupational Performance Measure (COPM) | For Group1: Change from pre-test at Day 1 (prior to training) to post-test 1 at Day 2. For Group 2: Change from pre-test 2 at Days 4-6 to post-test 1 at Days 5-7.
  COPM is an evidence-based outcome measure designed to capture a patient's self-perception of performance in everyday living (Law et al., 1994). One to five activities will be chosen by the participant. Range of possible scores is 1 [poor performance and low satisfaction] - 10 [very good performance and high satisfaction] per activity.
Mean somatosensory-evoked potential (SEP) latencies for N20 and N30 | For Group1: Change from pre-test at Day 1 (prior to training) to post-test 1 at Day 2. For Group 2: Change from pre-test 2 at Days 4-6 to post-test 1 at Days 5-7.
  SEPs after median nerve stimulation are recorded. The latencies for N20 and N30 will be identified. Unit is in milliseconds.
Peak-to-peak amplitude of motor-evoked potential (MEP) | For Group1: Change from pre-test at Day 1 (prior to training) to post-test 1 at Day 2. For Group 2: Change from pre-test 2 at Days 4-6 to post-test 1 at Days 5-7.
  Single-pulse transcranial magnetic stimulation (TMS) is used to assess corticospinal excitability by eliciting MEP of the wrist extensor muscles using a method described by Samargia et al. (2014). Unit is millivolts.

OTHER OUTCOMES:
Tactile sensitivity | Measured on the first day of the intervention
  Forearm tactile sensitivity assessment using the Semmes-Weinstein Monofilaments (Bell-Krotoski et al., 1995). Monfilaments measure both diminishing and returning cutaneous sensation. The monofilament bends at a force of 0.1N. Patient will report, yes, if the monofilament is perceived at that force level. Range of scores are + [perceived] and - [not perceived].

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Konczak, Ph.D, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Beck, A. T., Steer, R. A., & Carbin, M. G. (1988). Psychometric properties of the Beck Depression Inventory: Twenty-five years of evaluation. Clinical psychology review, 8(1), 77-100.
- [Background] Bell-Krotoski JA, Fess EE, Figarola JH, Hiltz D. Threshold detection and Semmes-Weinstein monofilaments. J Hand Ther. 1995 Apr-Jun;8(2):155-62. doi: 10.1016/s0894-1130(12)80314-0. PMID 7550627
- [Background] Folstein MF, Robins LN, Helzer JE. The Mini-Mental State Examination. Arch Gen Psychiatry. 1983 Jul;40(7):812. doi: 10.1001/archpsyc.1983.01790060110016. No abstract available. PMID 6860082
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Hislop, H., Avers, D., & Brown, M. (2013). Daniels and Worthingham's muscle testing: Techniques of manual examination and performance testing: Elsevier Health Sciences.
- [Background] Law M, Polatajko H, Pollock N, McColl MA, Carswell A, Baptiste S. Pilot testing of the Canadian Occupational Performance Measure: clinical and measurement issues. Can J Occup Ther. 1994 Oct;61(4):191-7. doi: 10.1177/000841749406100403. PMID 10137673
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Samargia S, Schmidt R, Kimberley TJ. Shortened cortical silent period in adductor spasmodic dysphonia: evidence for widespread cortical excitability. Neurosci Lett. 2014 Feb 7;560:12-5. doi: 10.1016/j.neulet.2013.12.007. Epub 2013 Dec 12. PMID 24333913
- [Background] Stolk-Hornsveld F, Crow JL, Hendriks EP, van der Baan R, Harmeling-van der Wel BC. The Erasmus MC modifications to the (revised) Nottingham Sensory Assessment: a reliable somatosensory assessment measure for patients with intracranial disorders. Clin Rehabil. 2006 Feb;20(2):160-72. doi: 10.1191/0269215506cr932oa. PMID 16541937
- [Background] Turgut N, Altun BU. Cortical disinhibition in diabetic patients with neuropathic pain. Acta Neurol Scand. 2009 Dec;120(6):383-8. doi: 10.1111/j.1600-0404.2009.01235.x. PMID 19922582
- [Derived] Yeh IL, Holst-Wolf J, Elangovan N, Cuppone AV, Lakshminarayan K, Cappello L, Masia L, Konczak J. Effects of a robot-aided somatosensory training on proprioception and motor function in stroke survivors. J Neuroeng Rehabil. 2021 May 10;18(1):77. doi: 10.1186/s12984-021-00871-x. PMID 33971912